CLINICAL TRIAL: NCT04060498
Title: Effectiveness of Mindfulness Intervention in Prevention of Relapse in Psychosis
Brief Title: Mindfulness Intervention and Relapse in Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: University Grants Committee, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17110918
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Psychosis
Keywords: Mindfulness, Prevention, Relapse, Psychosis, Schizophrenia, Psychotic Disorders, Mental Disorders, Schizophrenia and Disorders with Psychotic Features
MeSH Terms: conditions — Psychotic Disorders; Recurrence; Schizophrenia; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness intervention (Experimental): This arm consists of seven weekly-session mindfulness-based intervention for psychosis (MBI-p). The MBI-p is a protocol-based, low intensity intervention developed to help patients achieve a greater sense of peace and calmness, and facilitates participants in handling everyday stress and conflicts.
  Interventions: Behavioral: Mindfulness intervention
- Psychoeducation intervention (Placebo Comparator): This arm consists of seven weekly-sessions of psychoeducation. Topics to be discussed in the sessions include the signs and symptoms of psychosis, aetiology of psychosis, as well as pharmacological and non-pharmacological interventions.
  Interventions: Behavioral: Psychoeducation intervention

INTERVENTIONS:
Behavioral: Mindfulness intervention — MBI-p focuses on simplicity, for both facilitators and patients; and use acceptance and embracing attitude for fear and sadness. The ultimate aims are to help patients achieve a greater sense of peace and calmness, and facilitate participants in handling everyday stress and conflicts.
  Arms: Mindfulness intervention
Behavioral: Psychoeducation intervention — Psychoeducation focuses on disseminating information about common mental disorders, psychosis (its causes, risk factors and trajectory), and methods of treatment for psychosis.
  Arms: Psychoeducation intervention

SUMMARY:
Practicing mindfulness is popular and well-accepted for its benefits in improving mental and physical health. In particular, its benefits in promoting resilience to stress and well-being have been shown in studies involving different psychiatric conditions, as well as preventing relapse in patients with depressive disorders. However, its role in relapse prevention among patients with psychosis has not been tested.

The investigators therefore propose a multi-site, single-blind, 12-month randomized controlled trial in Hong Kong to examine the effectiveness of mindfulness intervention in prevention of relapse among 152 remitted psychosis patients.

DETAILED DESCRIPTION:
Objectives and hypotheses

1. Primary objective:

   • To examine if mindfulness-based intervention can reduce rates of relapse at 1 year in remitted patients with psychosis.
2. Secondary objectives:

   * To test whether mindfulness-based intervention can reduce stress, depressive symptoms, and improve functioning and quality of life at 1 year in remitted patients with psychosis.

Participants Patients will be recruited from the Early Assessment Service for Young people with psychosis (EASY). This service provides specialized psychiatric care for the first three years for young persons with first episode psychosis and covers the entire population of Hong Kong of approximately seven million people. The sample will consist of 152 fully remitted patients diagnosed with schizophrenia or non-affective psychosis (schizophreniform disorder, schizoaffective disorder, brief psychotic disorder, or psychotic disorder not otherwise specified)

Study design This is a single-blind, 12-month, multi-site, randomized controlled trial (RCT) of the effect of mindfulness intervention in preventing relapse in remitted psychosis. Patients will be randomized into either having 7-week mindfulness-based intervention or 7-week psychoeducation groups. The study consists of the following time points: baseline (before the start of intervention), at 7-week after the intervention, and then monthly for the remaining 12 months following end of the intervention. Relapse will be assessed monthly during the 1-year follow-up period. Patients will be terminated from the study if relapse occurs during the follow up. The study will be carried out in accordance with Good Clinical Practice and with the Declaration of Helsinki. The study have sought for approval from the Institutional Review Boards at each site. All participants will be required to provide written informed consent. Patients will be individually randomized to one of the two parallel groups: 7-week mindfulness intervention or 7-week psychoeducation.

Procedures

Mindfulness intervention group All patients in the mindfulness group will receive EASY service and 7 weekly-session mindfulness-based intervention for psychosis (MBI-p). It is a protocol-based, low intensity mindfulness developed to help patients to achieve greater sense of peace and calmness, and facilitate participants in handling everyday stress and conflicts. MBI-p consists of seven 1.5-hour group sessions, and each group will have 2-6 participants. Each MBI-p session has the following components: engagement and introduction, mindfulness practices, daily life application and consolidation of learning. Facilitators in conducting the MBI-p will be trained by experienced investigators.

Psychoeducation group All patients in the psychoeducation group will receive EASY service and 7 weekly-session psychoeducation. Each psychoeducation will last for 1.5 hours, including topics on the signs and symptoms of psychosis, aetiology of psychosis and medication usage.

Assessments The primary outcome of relapse will be assessed using the Positive and Negative Syndrome Scale (PANSS) and the Clinical Global Impressions (CGI) Scale (Guy, 1976). Relapse will be assessed before (baseline) and after intervention, and then monthly for 12 months. When patients experience a psychotic relapse at any point during this 12-month period, their participation will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 55 years
* in full symptomatic remission for at least 6 months
* have been ill for no more than 3 years following first episode psychosis
* have sufficient proficiency in Chinese to understand verbal instructions and to give informed consent.

Exclusion Criteria:

* known diagnosis of intellectual disability
* organic brain disorder
* current or previous use of illicit drugs
* substance-induced psychosis or alcohol intake in excess of 5 standard units per day
* people who practice mindfulness and meditation exercise for more than twice a week over the past 1 month.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with psychotic relapse(s) | 12 months post-intervention
  Psychotic relapse is defined as an increase in at least one of the following PANSS (Kay et al., 1987) items: delusion and/or hallucinatory behavior to a score of 3 or above; conceptual disorganization or unusual thought content to a score of 4 or above; and suspiciousness to a score of 5 or above.

CONTACTS AND LOCATIONS:
Overall Officials: Christy Lai-ming Hui, Dr, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guy W (1976). Clinical global impression scale (CGI). In Guy W. editors. ECDEU assessment manual for psychopharmacology, Revised. Rockville MD: US Dept of Health, Education and Welfare, National Institute of Mental Health. Page 217-222.
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518
- [Derived] Hui CLM, Wong CCL, Lui ECY, Chiu TC, Tao TJ, Chan EWT, Lin J, Tong ACY, Suen YN, Chan CWH, Yeung WS, Lee EHM, Chan SKW, Chang WC, Chen EYH. Effects of mindfulness-based intervention in preventing relapse in patients with remitted psychosis: a randomized controlled trial. Schizophrenia (Heidelb). 2024 Dec 20;10(1):120. doi: 10.1038/s41537-024-00539-0. PMID 39702769